CLINICAL TRIAL: NCT02026050
Title: Phase 4 Study of Comparison of Postoperative Analgesic Effect of Intra-articular Dexamethasone and Dexamethasone Added to Bupivacaine in Interscalene Brachial Plexus Blockade for Arthroscopic Shoulder Surgery
Brief Title: Analgesic Effect of Intra-articular Dexamethasone and Dexamethasone Added to Bupivacaine in Interscalene Brachial Plexus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Fatih Mehmet Kurt, resident, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013/639
Record Dates: First submitted 2013-12-30; First posted 2014-01-01 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Postoperative Pain
Keywords: dexamethasone; intraarticular injection; interscalene brachial plexus block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- intraarticular dexamethasone (Active Comparator): interscalene brachial plexus block was preoperative performed 30 ml 0.5 % bupivacaine+ 2 ml serum phsyologic and after surgery 2 ml 8 mg dexamethasone+ 8 ml serum phsyologic administration for intraarticular
  Interventions: Procedure: intraarticular dexamethasone
- interscalene dexamethasone (Active Comparator): interscalene brachial plexus was preoperative performed 30 ml 0.5 % bupivacaine added 2 ml 8mg dexamethasone and after surgery 10 ml serum phsyologic administration for intraarticular
  Interventions: Procedure: interscalene dexamethasone
- serum phsyologic (Placebo Comparator): interscalene brachial plexus block was preoperative performed 30 ml 0.5 % bupivacaine+ 2ml serum phsyologic and after surgery 10 ml serum phsyologic administration for intraarticular
  Interventions: Procedure: serum phsyologic

INTERVENTIONS:
Procedure: intraarticular dexamethasone — 2ml 8 mg dexamethasone administration for intraarticular
  Other Names: dekort
  Arms: intraarticular dexamethasone
Procedure: interscalene dexamethasone — 2ml 8 mg dexamethasone administration interscalene brachial plexus added 30 ml 0.5 % bupivacaine
  Other Names: dekort
  Arms: interscalene dexamethasone
Procedure: serum phsyologic — interscalene brachial plexus block was preoperative performed 30 ml 0.5 % bupivacaine+ 2ml serum phsyologic and after surgery 10 ml serum phsyologic administration for intraarticular
  Arms: serum phsyologic

SUMMARY:
the aim of this study was to investigate the analgesic efficacy of intra articular dexamethasone administration for arthroscopic shoulder surgery.

DETAILED DESCRIPTION:
shoulder surgery can be very painful and interscalene brachial plexus block is the gold standard in the management of acute pain after shoulder surgery. various local anaesthetic mixtures can be used to prolong local anaesthesia duration and epinephrine , opioids and dexamethasone are frequently used for this purpose. dexamethasone has also been found the prolong the duration of lidocaine axillary blocks and intravenous regional anaesthesia. intraarticular administration of medicines can be used for management of joint pain and opioids , local anaesthetics and dexamethasone are used for this purpose.In addition, there are no studies available to compare the different treatment methods used in clinical practice directly.

ELIGIBILITY:
Inclusion Criteria:

* between 18-65 years
* arthroscopic shoulder surgery
* no known allergies to drugs
* ASA 1-2 patients

Exclusion Criteria:

* history of diabetes
* history of chronic pain treatment
* pregnancy
* severe bronchopulmonary disease
* systemic glucocorticoid use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2014-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
analgesic consumption | postoperative 1 day
  morphine consumption (patient controlled analgesia procedure) was recorded

SECONDARY OUTCOMES:
visual analog scale | postoperative 1 day
  Visual analog scale on rest and movement was recorded

CONTACTS AND LOCATIONS:
Overall Officials: Fatih M KURT, Resident, Principal Investigator — TC Erciyes University; Gülen GÜLER, Prof., Study Director — TC Erciyes University
Locations (1):
- Erciyes university hospital, Kayseri, Turkey (Türkiye)